CLINICAL TRIAL: NCT04900064
Title: Evaluation of Primary Care Behavioral Health (PCBH) With the Addition of Self-help CBT - A Randomized Multicenter Trial for Superiority and Non-superiority Comparisons of Effects on Patients' Everyday Function, Symptoms, and Experiences
Brief Title: Evaluation of Primary Care Behavioral Health (PCBH) With the Addition of Self-help CBT - A Randomized Multicenter Trial
Acronym: KAIROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other); Capio Group (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-04198-A2
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Panic Disorder; Social Anxiety Disorder; Depression; Hypochondriasis; Insomnia; Generalized Anxiety Disorder; Burnout; Adjustment Disorders; Stress, Psychological; Obsessive-Compulsive Disorder; Life Stress; Life Style Induced Illness; Psychological Distress
MeSH Terms: conditions — Panic Disorder; Phobia, Social; Depression; Hypochondriasis; Sleep Initiation and Maintenance Disorders; Generalized Anxiety Disorder; Burnout, Psychological; Adjustment Disorders; Stress, Psychological; Obsessive-Compulsive Disorder | interventions — Crisis Intervention; Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Patients are randomised between a diagnostic assessment and a contextual assessment. Patients in the contextual assessment arm can only be treated with brief interventions whereas patients in the diagnostic assessment arm are offered guided self-help if deemed appropriate and otherwise gets brief interventions.
  As such, patients are randomised between two arms. We have however included four arms below in order to be able to describe the primary and secondary analysis. The primary analysis is performed on all patients treated with self-help CBT in the arm where a diagnostic assessment is made, compared to patients in the contextual assessment arm that are found suitable for self-help CBT (based on screening data), but treated with brief interventions.
Who Masked: Participant
Masking Description: Patients will only be informed that they will be randomised between two different types of extended assessments, both of which are more extensive than regular healthcare. They will receive no information about the nature of the assessments or about different treatments following the assessments to avoid nocebo effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diagnostic Assessment - Given self-help CBT (Experimental): The diagnostic assessment includes screening instruments, a structured interpretation of the screening instruments, a structured interview (MINI - International Neuropsychiatric Interview) and a medical anamnesis. If deemed appropriate, the patient can be offered treatment with guided self help. If the patient's problem is not deemed appropriate for this type of care or if the patient is not interested in guided self-help, they are offered brief interventions (BI).
  In the primary analysis, only patients receiving treatment with self-help CBT are included.
  Interventions: Behavioral: Self-help CBT
- Contextual Assessment - Suitable for self-help CBT but given brief interventions (Active Comparator): The contextual assessment includes screening instruments and a contextual interview. Patients in this arm will always be treated with brief interventions.
  In the primary analysis, only patients suitable for self-help CBT are included. This is decided by an algorithm based on data from their screening, which takes into account symptom severity and type, patient preference and known variables that make self-help CBT a worse fit.
  Interventions: Behavioral: Brief interventions
- Diagnostic Assessment - All patients (Experimental): Same as the other arm marked as "Experimental", but for the purpose of a secondary analysis all patients randomised to Diagnostic Assessment are included, regardless if they receive treatment with self-help CBT or brief interventions.
  Interventions: Behavioral: Brief interventions; Behavioral: Self-help CBT
- Contextual Assessment - All patients (Active Comparator): Same as the other arm marked as "Experimental", but for the purpose of a secondary analysis all patients randomised to Diagnostic Assessment are included, regardless if they are deemed suitable for self-help CBT or not.
  Interventions: Behavioral: Brief interventions

INTERVENTIONS:
Behavioral: Brief interventions — 'Brief Interventions' (BI) is a generic term for a multitude of tools and interventions used in patient visits within PCBH. BI start immediately at the initial consultation, which ends with a personally tailored and evidence-informed plan adjusted to the patient's context. As such, there is no separation between assessment and intervention. The interventions within BI often have their foundation in CBT, ACT or Motivational Interviewing (MI). The common theme is that they are principle-based rather than manual-based and focus on behavioural change in relation to a problem, rather than focusing on a specific diagnosis. Follow-up appointments are scheduled flexibly depending on the patient's perceived need. A BI treatment usually consists of 1-4 appointments with several weeks apart and has an open ending, where the patient easily can schedule a new appointment. Clinicians delivering brief interventions will have had 3 days of training as well as regular supervision.
  Other Names: Focused CBT, focused ACT, Focused Cognitive Behavioural Therapy, Focused Acceptance and Commitment Therapy
  Arms: Contextual Assessment - All patients; Contextual Assessment - Suitable for self-help CBT but given brief interventions; Diagnostic Assessment - All patients
Behavioral: Self-help CBT — The patient receives a previously scientifically evaluated CBT-based self-help book for one of the following conditions: depression, generalized anxiety disorder, panic disorder, social anxiety, health anxiety, insomnia, or stress/burnout. The therapist support consists of 3-6 contacts throughout the 6-12 weeks long intervention period as decided by the clinician and patient together, as long as at least one and not more than three are physical visits at the center and the rest via phone, video conferencing, or secure internet messages. Clinicians delivering self-help CBT will need four days of reading and two days of training as well as regular supervision to be able to make initial assessments and problem profiling and use the self-help books.
  Other Names: Bibliotherapy, iCBT, Internet-Based Cognitive Behavioural Therapy, Blended Treatment, Self-help books
  Arms: Diagnostic Assessment - All patients; Diagnostic Assessment - Given self-help CBT

SUMMARY:
In this multicenter study, the investigators want to find out if an addition of an diagnostic assessment and possibility of treatment with guided self-help CBT can increase the treatment effects of PCBH on patient functioning and symptoms, compared to standard PCBH which uses contextual assessment and brief interventions. In addition to this, the study will investigate the overall effect of PCBH on both patient and organisation level outcomes.

DETAILED DESCRIPTION:
The overarching goal of primary care is to offer all patients individualised and context-sensitive healthcare with high access and continuity. One of the reasons primary care struggles with this goal is that a large proportion of patients suffer from mental and behavioural health problems, alone or in combination with one or several chronic illnesses. Despite many patients needing psychosocial interventions, there is a lack of mental health professionals as well as clear pathways for these patients.

Primary Care Behavioural Health (PCBH) is an innovative way of organising primary care, where mental health professionals have more yet shorter visits, strive for same-day access, and have an active consulting role in the primary care team. To help patients achieve relevant behavioural changes, so called brief interventions are used, which are based on isolated components from psychological treatments such as Cognitive Behavioural Therapy (CBT) and Acceptance and Commitment Therapy (ACT). Brief interventions usually stretch over 1-4 treatment sessions. Assessments within the model are generally contextual and largely avoid psychiatric diagnostics, instead focussing on the patient's situation and their associated coping strategies - whether they be positive or negative. However, these interventions have not been systematically evaluated in the same way that structured CBT has, and there is a risk that patients that would have benefitted from structured CBT and a diagnostic assessment are undertreated due to lack of diagnostics and the reduced visit duration and amount.

Data will be collected at primary care centres (PCCs) that already have a high fidelity to a PCBH framework. Fidelity will be measured by an expert group as well as using four questionnaires, one for each of mental health professionals, medical doctors, registered nurses and leadership. These fidelity scales will be validated in a separate study. In addition to fidelity, work environment and satisfaction with the PCBH implementation will be measured.

Patients at the centres will be randomised between receiving contextual assessments followed by brief interventions, or a diagnostic assessment, which can lead to treatment with either self-help CBT (if a treatable diagnosis is confirmed and the patient is suitable for self-help CBT) or brief interventions (if self-help CBT is not deemed to be a suitable intervention). The primary comparison is the outcome for patients who either received self-help CBT or are deemed suitable for the intervention based on screening data, while secondary analyses will look at treatment outcomes for all patients, including those with non-psychiatric problems such as crises, loss or work- or family-related problems. The study will also look at implementation outcomes for self-help CBT and diagnostic assessments to see if self-help CBT is a feasible addition to the PCBH model. Our main research questions are:

1. Does an extended version of PCBH, including an additional assessment and the option of guided self-help CBT when indicated by a patient's problem profile, lead to superior patient outcomes compared to standard PCBH where a brief, contextual assessment followed by Brief Interventions is the only option? If not, can standard PCBH be shown to be non-inferior?
2. Does the addition of guided self-help CBT have a negative effect on availability, reach, and cost-effectiveness compared to standard PCBH? If not, can guided self-help CBT be shown to be non-inferior to standard PCBH concerning these outcomes?

PCBH has the potential to increase the quality and access of care for many patients with mental and behavioural health problems. This study is the first to step towards answering whether or not the effects of brief intervention are large enough to merit large-scale implementation, and if an add-on of other brief and easily implementable treatments can increase the treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* All patients from age 18 who seek care at the PCC, who are deemed to be suitable for Behavioural Health interventions and booked to the mental health professionals at the PCC, according to screening methods and/or clinical assessments made by health care personnel at the PCC, will be included. This broad criteria reflects the naturalistic setting where decisions of clinicians, rather than highly standardized criteria, are the basis for inclusion.

Exclusion Criteria:

* Does not speak Swedish well enough to fill out questionnaires or to receive self-help CBT in Swedish.
* Is in need of emergency type care, like with suicidal ideation or behaviours, ongoing psychosis or mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1242 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
WHO Disability Assessment Schedule 2.0 12-item (WHODAS-12) (4 domains) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  The four domains of Life activities, Cognition, Getting along, and Participation. In the 12-item version of the WHO Disability Assessment Schedule 2.0 (WHODAS-12) will be used as primary outcome, since these are condition-independent measures of Behavioral Health relevant everyday functioning. The scale ranges from 0 to 32 points. A lower score means better functioning. As such, a lower score is a better outcome.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule 2.0 12-item (WHODAS-12) (whole instrument) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  The two domains of Mobility and Self-care will be measured and the whole WHODAS will be used in some secondary analyses, but not for the primary outcome since these domains tend to form two independent factors, many patients will have initial adequate function in these domains and they are not expected to change much. The scale ranges from 0 to 48 points. A lower score means better functioning. As such, a lower score is a better outcome.
Patient Health Questionnaire 9-Item (PHQ-9) | Change during the period Pre, Week 12 and 1 year
  The full version of a well-validated scale for measuring depressive symptoms. PHQ-9 total score for the nine items ranges from 0 to 27. A lower score means less depressive symptoms. As such, a lower score is a better outcome.
Patient Health Questionnaire 2-Item (PHQ-9) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  PHQ-2 consists of two questions from the PHQ-9. This will be administered as part of the PHQ-9 on the above mentioned time points, and will replace the PHQ-9 on the mid-treatment measurements. The scale ranges from 0 to 6 points. A lower score means less depressive symptoms. As such, a lower score is a better outcome.
Generalized Anxiety Disorder 7-item (GAD-7) | Change during the period Pre, Week 12 and 1 year
  The full version of a well-validated scale for measuring anxiety symptoms. GAD-7 total score for the seven items ranges from 0 to 21. A lower score means less anxiety symptoms. As such, a lower score is a better outcome.
Generalized Anxiety Disorder 2-item (GAD-2) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  GAD-2 consists of two questions from the GAD-7. This will be administered as part of the GAD-7 on the above mentioned time points, and will replace the GAD-7 on the mid-treatment measurements. The scale ranges from 0 to 6 points. A lower score means less anxiety symptoms. As such, a lower score is a better outcome.
Social Phobia Inventory - Abbreviated version (Mini-SPIN) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Social anxiety symptoms are measured with a very short version of a well established patient-rated scale for social phobia. The scale ranges from 0 to 12 points. A lower score means less symptoms of social anxiety. As such, a lower score is a better outcome.
The Alcohol Use Disorders Identification Test-Concise (AUDIT-C) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of alcohol misuse are measured with a very short version of a well established patient-rated scale for alcohol misuse. The scale ranges from 0 to 12 points. A lower score means less symptoms of alcohol misuse. As such, a lower score is a better outcome.
Panic Disorder Severity Scale - Self rated 2-item (PDSS-SR-MINI-2) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of panic attacks are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 8 points. A lower score means less symptoms of panic disorder. As such, a lower score is a better outcome.
Karolinska Exhaustion Disorder Scale 3-item (KEDS-3) + 2 confirming questions from s-UMS | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of stress-related exhaustion are measured with a very short version of a well established patient-rated scale and has been created by an expert group, who chose three representative questions from the original KEDS scale. To aid with diagnostics, two confirmatory questions from the Swedish s-UMS scale were added, asking for duration and presumed cause of symptoms. The scale ranges from 0 to 18 points. A lower score means less symptoms of stress-related exhaustion. As such, a lower score is a better outcome.
Perceived Stress Scale (PSS-MINI-2) + 2 new questions | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Stress symptoms are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. To increase face validity of the very short scale, we also added two more direct questions ("Have you been feeling stressed lately?", "Have you been feeling tense lately?"). The scale ranges from 0 to 16 points. A lower score means less stress symptoms. As such, a lower score is a better outcome.
Insomnia Severity Index 2-item (ISI-MINI-2) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of sleep disorders are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 8 points. A lower score means less sleep problems. As such, a lower score is a better outcome.
Short Health Anxiety Inventory 3-item (SHAI-MINI-3) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of health anxiety are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 9 points. A lower score means less symptoms of health anxiety. As such, a lower score is a better outcome.
Obsessive Compulsive Disorder 3-Item (OCD-3-MINI) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Symptoms of obsessive compulsive disorder are measured by a very short patient-rated scale and has been created by an expert group. The scale ranges from 0 to 12 points. A lower score means less obsessive/compulsive thoughts and behaviors. As such, a lower score is a better outcome.
Pain One-item Rating | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Pain is measured on a scale from 0 to 10, where 0 is no pain and 10 is worst pain imaginable. As such, a lower score is a better outcome.
Total symptom index | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  Also, a total index for level of symptoms will be calculated from all symptom items, where different weights will be used to balance the different number of questions for different domains, for example to avoid the larger number of items related to anxiety to overshadow depression ratings. The scale ranges from 0 to 20 points. A lower score means less mental health symptoms overall. As such, a lower score is a better outcome.
Brunnsviken Brief Quality of Life Questionnaire (BBQ) | Change during the period Pre, Week 12 and 1 year
  Quality of life will be measure be the 12-item Brunnsviken Brief Quality of life (BBQ-12), asking about importance and fulfilment of six areas (e.g. spare time quality, creative work, and friendship). The scale ranges from 0 to 96 points. A lower score means lower quality of life. As such, a higher score is a better outcome.
Outcome Rating Scale (ORS) | Change during the period Pre, Week 4, Week 8, Week 12 and 1 year
  The ORS is a four-item measure designed to assess areas of life functioning known to change as a result of therapeutic intervention. These include symptom distress, interpersonal well-being, social role, and overall well-being, measured by four visual analogue scales. The scale ranges from 0 to 40 points. A lower score means lower satisfaction with life areas. As such, a higher score is a better outcome.
Session Rating Scale (SRS) | Week 4, Week 8, Week 12 and 1 year
  The Session Rating Scale (SRS) is a four-item visual analogue scale designed to assess key dimensions of effective therapeutic relationships. These include respect and understanding, relevance of the goals and topics, client-practitioner fit and overall alliance. The scale ranges from 0 to 40 points. A lower score means lower ratings of the therapeutic alliance. As such, a higher score is a better outcome.
One item Clinical Global Impression - Improvement (CGI-I) | After every session during week 1-12
  Related to main problem seeking care for as rated by clinician. The scale ranges from 0 to 7 points. A lower score means a larger improvement for the patient. As such, a lower score is a better outcome.
Patient-rated perception and attitude toward care provider | Week 12
  9-items previously used in PCBH-settings (self-report), and four items from the Client Satisfaction Questionnaire (CSQ). The scale ranges from 0 to 57 points. A lower score means less satisfaction with care. As such, a higher score is a better outcome.
Description of Behavioral Health Plan (PCBH) or main treatment goal and methods (shCBT) as structured note by clinician in medical record | Week 12
  Interview form.
Patient recollection of plan/goal/methods, descriptions of behaviour changes made | Week 12
  Interview form.
Experienced negative/Adverse Events, where the worst and most probably care-induced event is more thoroughly described and rated on severity and perceived cause | Week 12
  Interview form.
Adverse Events-9 | Week 12
  9 items asking patients to detail any adverse events that occurred as a result of treatment.
Adverse Events-3 | Week 4, Week 8
  3 items asking patients to detail any adverse events that occurred as a result of treatment.
Well-being Behaviours-11 | Change during the period Pre, Week 12 and 1 year
  11 items asking patients how often they engage in behaviours related to maintaining physical and mental well-being, such as physical exercise and having adequate sleep hygiene.

OTHER OUTCOMES:
Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Pre, Week 12, 1 year
  The TIC-P is a validated patient-reported outcome measure concerning the utilization of medical care and productivity losses. It does not have a minimum or maximum score but collects information that is needed for doing health economic calculations. This includes outcome measures such as amount of days on sick leave, productivity loss when at work, productivity loss at home, and medications prescribed and taken. Patient self-report will be complemented with register-level data on sick leave and medications.
Average waiting time | At first visit
  - Average waiting time from the identification of a behavioural health concern to being seen by any clinician among patients in the study
Supply of bookable appointments | Weekly from study start up to 2 years
  Amount of bookable times per week and full time psychosocial resources (personnel in training counted as 75% of full time), an indirect measure of availability to psychosocial resources
Third next available appointment (TNAA) | Weekly from study start up to 2 years
  Waiting time until next available appointment for a third hypothetical patient that calls in on a given day for every clinician at the PCC, measured on the same time every week (e. g. Mondays at 9 AM), a measure of access to and and availability of care
Future capacity | Weekly from study start up to 2 years
  Number of available time slots for appointments in the coming 4 weeks divided by total number of time slots in the caregiver's calendar, an indirect measure of availability
Number of visits and phone / video contacts during treatment duration | All visits during Pre-Week 12
  Average number of visits per treatment, averaged across groups
Average visit length | All visits during Pre-Week 12
  Average length of visits with psychosocial resources, averaged across groups
Percentage of patients presenting with a new primary reason for visit or more than 6 months since last visit | Daily from study start up to 2 years
  An indirect measure of reach of psychosocial interventions
The number of patients seen per full time equivalent mental health professional for at least one visit in relation to all patients listed at the PCC | Monthly from study start up to 2 years
  A measure of reach of psychosocial interventions
The number of patients seen per full time equivalent mental health professional for at least one visit in relation to all patients with an ICD-10 diagnosis of F10-99, R40-45 or Z55-65 | Monthly from study start up to 2 years
  A measure of reach of psychosocial interventions
Integrated Behaviours in Primary Care - Psychosocial Resource Edition (IBPC-PSR) | Pre, 6 months, 1 year
  To measure PCBH fidelity and competence among psychosocial resources
  This questionnaire is not yet validated and has been created by the research group, as previously existing questionnaires have been difficult to apply to the Swedish healthcare system. The questionnaires will be validated parallel to this study. The scales include subscales to measure several specific areas of interest, such as collaboration between psychosocial resources and medical personnel.
Levels of Integration Measure, Swedish version (S-LIM) | Pre, 6 months, 1 year
  To measure PCBH fidelity and competence among leaders
  This questionnaire is not yet validated and has been created by the research group, as previously existing questionnaires have been difficult to apply to the Swedish healthcare system. The questionnaires will be validated parallel to this study. The scales include subscales to measure several specific areas of interest, such as collaboration between psychosocial resources and medical personnel.
Integrated Behaviours in Primary Care - Registered Nurse Edition (IBPC-RN) | Pre, 6 months, 1 year
  To measure PCBH fidelity and competence among nurses
  This questionnaire is not yet validated and has been created by the research group, as previously existing questionnaires have been difficult to apply to the Swedish healthcare system. The questionnaires will be validated parallel to this study. The scales include subscales to measure several specific areas of interest, such as collaboration between psychosocial resources and medical personnel.
Integrated Behaviours in Primary Care - GP Edition (IBPC-GP) | Pre, 6 months, 1 year
  To measure PCBH fidelity and competence among doctors
  This questionnaire is not yet validated and has been created by the research group, as previously existing questionnaires have been difficult to apply to the Swedish healthcare system. The questionnaires will be validated parallel to this study. The scales include subscales to measure several specific areas of interest, such as collaboration between psychosocial resources and medical personnel.
Self-help CBT fidelity | Pre, 6 months, 1 year
  11 questions created by an expert group measuring fidelity to self-help CBT treatment.
Attitudes to brief interventions | Pre, 6 months, 1 year
  The AIM-IAM-FIM measurement with the three subscales Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM) to measure implementation constructs acceptability, appropriateness and feasibility of PCBH implementation
Attitudes to self-help CBT | Pre, 6 months, 1 year
  The AIM-IAM-FIM measurement with the three subscales Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM) to measure implementation constructs acceptability, appropriateness and feasibility of self-help CBT implementation
Implementation success of PCBH | Pre, 6 months, 1 year
  The original British instrument the Normalization Process Theory Measure (NoMAD) is based on the four core constructs of the Normalization Process Theory: Coherence, Cognitive Participation, Collective Action, and Reflexive Monitoring. They represent ways of thinking about implementation and are focused on how interventions can become part of everyday practice. The s-NoMAD is the validated Swedish version of the NoMAD.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Professor, Principal Investigator — Linnaeus University, Karolinska Institutet
Locations (4):
- Sweden (4):
  - Vårdcentralen Västra Vall, Varberg, Halland County
  - Capio Citykliniken Västra Hamnen, Malmo, Skåne County
  - Boo vårdcentral, Stockholm, Stockholm County
  - Capio Vårdcentral Sävja, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farnsworth von Cederwald A, Salomonsson S, Hentati Isacsson N, Kaldo V. Evaluation of Primary Care Behavioral Health (PCBH) with guided self-help CBT as a treatment option - a protocol of a single-blind randomized multicenter trial (KAIROS). BMC Health Serv Res. 2025 Sep 23;25(1):1208. doi: 10.1186/s12913-025-13232-4. PMID 40988013